CLINICAL TRIAL: NCT04725227
Title: Determine the Effect of Prone Positioning on Lung Ventilation and Perfusion Distribution in Adults With Acute Respiratory Distress Syndrome by Electrical Impedance Tomography
Brief Title: Determine the Effect of Prone Positioning in Adults With ARDS by Electrical Impedance Tomography
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Principal Investigator, Ming Zhong, Professor, Shanghai Zhongshan Hospital
Other Study IDs: P-E
Record Dates: First submitted 2021-01-25; First posted 2021-01-26 (Actual); Last update posted 2021-01-26 (Actual); Status verified 2021-01

CONDITIONS: ARDS; Prone Position; Electrical Impedance Tomography

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
determine the effect of prone positioning on ventilation and perfusion distribution in adults with acute respiratory distress syndrome by electrical impedance tomography

DETAILED DESCRIPTION:
By intravenous injection of a small amount of normal saline, electrical impedance tomography enables evaluation of the pulmonary blood flow. EIT might be helpful in establishing the hypoxemia etiology at bedside via combining regional ventilation and perfusion information. The objective of this study was to describe the physiological effects of prone position on respiratory mechanics, ventilation and pulmonary perfusion in patients with ARDS.

ELIGIBILITY:
Inclusion Criteria:

* patients who were undergoing mechanical ventilation with moderate-to-severe ARDS (defined as a Pao2:Fio2 ratio < 150 mm Hg with a positive end-expiratory pressure ≥ 5 cm of water, and an Fio2 of ≥ 0.6) according to the Berlin definition

Exclusion Criteria:

* contraindications to the use of EIT (e.g., presence of pacemaker or chest surgical wounds dressing)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients requiring mechanical ventilation are recieved prone position ventilation who admitted to the surgical ICU.
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2020-12-01 (Actual); Primary Completion 2022-12-01 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Assess regional distribution of pulmonary perfusion | within 24 hours
  To evaluate the effect of prone positon on pulmonary blood flow distribution.
Assess regional distribution of pulmonary ventilation | within 24 hours
  To evaluate the effect of prone positon on pulmonary vetilation distribution.
Assess oxygenation status | within 24 hours
  To evaluate the effect of prone position by assessing regional distribution of pulmonary perfusion based on indicator dilution and changes at different points in time during varying states of regional ventilation will be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Ming Zhong, MD, phD, Principal Investigator — Fudan University
Locations (1):
- Zhongshan Hospital of Fudan University, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Wang Y, Muhetaer Y, Zheng X, Wu W, Tao J, Zhu L, Song J, Zhao Z, Zhong M. Time-dependent effects of prone position on ventilation-perfusion matching assessed by electrical impedance tomography in patients with COVID-19 ARDS: sub-analysis of a prospective physiological study. Ann Intensive Care. 2025 Mar 31;15(1):46. doi: 10.1186/s13613-025-01452-0. PMID 40163279
- [Derived] Wang Y, Song J, Lin S, Zheng X, Zhao Z, Zhong M. Influence of Prone Position on Regional Ventilation/Perfusion Matching in Patients With ARDS Over Time. Respir Care. 2025 Jul;70(7):821-829. doi: 10.1089/respcare.12247. Epub 2025 Mar 5. PMID 40040422
- [Derived] Wang YX, Zhong M, Dong MH, Song JQ, Zheng YJ, Wu W, Tao JL, Zhu L, Zheng X. Prone positioning improves ventilation-perfusion matching assessed by electrical impedance tomography in patients with ARDS: a prospective physiological study. Crit Care. 2022 May 27;26(1):154. doi: 10.1186/s13054-022-04021-0. PMID 35624489